CLINICAL TRIAL: NCT04589403
Title: A Phase 1a/1b Study of OPT101 in Healthy Volunteers
Brief Title: 1a/1b Study of OPT101 First in Human Study Assessing Safety and Tolerability of 15-mer Peptide.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Op-T LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: OPT-100-30
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Sentinel dosing of two subjects followed by review of the data by the Data Monitoring Committee (DMC) will be performed prior to enrolling any additional subjects within a cohort. Groups of 3 subjects (2 active:1 placebo) each will be treated at each dose level; for a total of 15 subjects. Additional subjects may be added to any cohort if dose limiting toxicity (DLT) is observed for a maximum of up to 6 subjects per cohort. An additional 6 subjects may also be enrolled in an intermediate dose cohort between the dose level which exceeds the defined MTD and the previous defined dose level.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Pharmacist will be the only unmasked clinical staff as the preparer of the investigational product prior to infusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.9% Sodium Chloride Injection USP (Placebo Comparator): Placebo will be 50 mL normal saline (Sodium Chloride), USP sterile solution administered by IV infusion over 30 minutes.
  Interventions: Drug: OPT101
- OPT101 (Experimental): The starting dose for the Phase 1a study is 0.16 mg/kg, which is 35-fold lower than the dog NOAEL (10mg/kg), on a mg/m2 basis. The dosing frequency for the MAD study was selected based on dosing performed in the supporting animal model studies. For an additional safety factor, the dose and volume infusion rates for the 0.16 mg/kg dose in humans will be 67-fold and 14-fold lower than the dogs dosed at 10mg/kg/min and mL/kg/min basis, respectively. For both Phase 1a and 1b, OPT101 will be administered by a slow IV infusion over 30 minutes.
  Interventions: Drug: OPT101

INTERVENTIONS:
Drug: OPT101 — 15-mer peptide with sequence based on the mouse CD154 domain interacting with CD40
  Other Names: 15-mer peptide

SUMMARY:
This is a first-in-human study, Phase 1, randomized, placebo-controlled, double blinded study that will be conducted in 2 parts.

DETAILED DESCRIPTION:
2 part study description:

• an initial Phase 1a single ascending dose (SAD) phase to identify a safe dose of OPT101.

Dose escalation will be by a factor of 2.6: 0.16, 0.42, 1.1, 2.8 and 7.3mg/kg.

• a Phase 1b multiple ascending dose (MAD) phase to measure safety and clinical effects of the highest and next to highest dose of OPT101 that are found to be safe in Phase 1a.

ELIGIBILITY:
Inclusion :

* Able and willing to give informed consent for the trial
* Male or female aged ≥18 years on the day of signing informed consent
* Is medically stable based on physical examination, medical history, laboratory results, and vital signs performed at screening
* Women of childbearing potential must have a negative highly sensitive serum test (beta-human chorionic gonadotropin) at screening and a negative urine pregnancy test at the Visit 1 Day 1 prior to receiving the investigational product.
* Women must agree to use one of the following methods of birth control for the duration of the clinical trial: systemic hormonal contraceptive (oral, injected, transdermal), intrauterine device, double barrier (e.g., cervical cap or diaphragm with condom or spermicide). Men with female partners must agree to use double barrier contraception, unless their partner is using systemic hormonal contraceptives or has an intrauterine device.

Exclusion:

* Is over the age of 55 years old
* Positive COVID test at screening/baseline
* Has an active fever or has recently been exposed to a COVID-19 patient.
* Currently has or had a history of malignancy
* Has an immune deficiency syndrome (for example, severe combined immunodeficiency syndrome, T-cell deficiency syndromes, B-cell deficiency syndromes, or chronic granulomatous disease), or bone marrow or organ transplantation, or a disease associated with lymphopenia
* Is currently being treated for an autoimmune disease/s
* Subjects with a history of venous and arterial thromboembolic events including, but not limited to, the following: deep venous thrombosis, pulmonary embolism, myocardial infarction, stroke, transient ischemic attack, or arterial insufficiency causing digital gangrene should be excluded. In addition, subjects with recent immobilization or recent surgery, should be excluded. Subjects with a history of abnormal prothrombotic laboratories such as congenital or inherited deficiency of antithrombin III, protein C, protein S, or confirmed diagnosis of antiphospholipid syndrome should also be excluded.
* Has active infections, is prone to infections or has chronic, recurrent or opportunistic infectious disease, including but not limited to, Epstein-Barr virus (EBV), cytomegalovirus (CMV) chronic renal infection, chronic chest infection, sinusitis, recurrent urinary tract infection, Pneumocystis carinii, aspergillosis, latent or active granulomatous infection, histoplasmosis, or coccidioidomycosis or an open, draining, or infected non-healing skin wound or ulcer
* Has recent or active hepatitis A infection, current/chronic hepatitis B and hepatitis C infection, or HIV infection. Participants with immunity to hepatitis B from previous infection (defined as negative HBsAg, positive anti-HBc, and positive hepatitis B surface antibody [anti-HBs]) or vaccination (defined as negative HBsAg, negative anti-HBc, and positive anti-HBs) may be eligible to participate.
* Has history of immune suppression disorders
* Has received a live (attenuated) vaccine within the last 60 days, including subjects who plan to receive live (attenuated) vaccines during the study or within 60 days after the final dose of study treatment.
* Has received influenza vaccine within 14 days of screening.
* Has received a biologic or immunotherapy in the last 6 months (If receiving allergy shots with stable dosing, is acceptable)
* Has received prescription or non-prescription medication and in the opinion of the Investigator, the product will interfere with the study procedures or data integrity or compromise the safety of the subject.
* Subjects with clinically significant abnormal laboratory test values in screening blood samples. In particular subjects with the following should be excluded:

Subjects with abnormal coagulation panel at screening such as abnormal PT or aPTT or fibrinogen

Abnormal liver function tests:

Liver enzyme abnormalities (except in the case of known Gilbert's syndrome) AST or ALT ≥3x ULN and total bilirubin ≥2x ULN AST or ALT ≥5x ULN AST or ALT ≥3x ULN if associated with appearance or worsening of rash or hepatitis symptoms Abnormal platelet counts (<150,000/mcL or > 450,000/mcL) Abnormal white blood cell counts (<3E3/uL or > 11E3/uL ) Abnormal eGFR (<60 mL/min/1.73m2) Elevated IgE level above 50 IU/mL

* Subjects planning to undergo Elective procedures or surgeries at any time after signing the ICF through the follow-up visit.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting withInclusion :
* Able and willing to give informed consent for the trial
* Male or female aged ≥18 years on the day of signing informed consent
* Is medically stable based on physical examination, medical history, laboratory results, and vital signs performed at screening
* Women of childbearing potential must have a negative highly sensitive serum test (beta-human chorionic gonadotropin) at screening and a negative urine pregnancy test at the Visit 1 Day 1 prior to receiving the investigational product.
* Women must agree to use one of the following methods of birth control for the duration of the clinical trial: systemic hormonal contraceptive (oral, injected, transdermal), intrauterine device, double barrier (e.g., cervical cap or diaphragm with condom or spermicide). Men with female partners must agree to use double barrier contraception, unless their partner is using systemic hormonal contraceptives or has an intrauterine device.

Exclusion:

* Is over the age of 55 years old
* Positive COVID test at screening/baseline
* Has an active fever or has recently been exposed to a COVID-19 patient.
* Currently has or had a history of malignancy
* Has an immune deficiency syndrome (for example, severe combined immunodeficiency syndrome, T-cell deficiency syndromes, B-cell deficiency syndromes, or chronic granulomatous disease), or bone marrow or organ transplantation, or a disease associated with lymphopenia
* Is currently being treated for an autoimmune disease/s
* Subjects with a history of venous and arterial thromboembolic events including, but not limited to, the following: deep venous thrombosis, pulmonary embolism, myocardial infarction, stroke, transient ischemic attack, or arterial insufficiency causing digital gangrene should be excluded. In addition, subjects with recent immobilization or recent surgery, should be excluded. Subjects with a history of abnormal prothrombotic laboratories such as congenital or inherited deficiency of antithrombin III, protein C, protein S, or confirmed diagnosis of antiphospholipid syndrome should also be excluded.
* Has active infections, is prone to infections or has chronic, recurrent or opportunistic infectious disease, including but not limited to, Epstein-Barr virus (EBV), cytomegalovirus (CMV) chronic renal infection, chronic chest infection, sinusitis, recurrent urinary tract infection, Pneumocystis carinii, aspergillosis, latent or active granulomatous infection, histoplasmosis, or coccidioidomycosis or an open, draining, or infected non-healing skin wound or ulcer
* Has recent or active hepatitis A infection, current/chronic hepatitis B and hepatitis C infection, or HIV infection. Participants with immunity to hepatitis B from previous infection (defined as negative HBsAg, positive anti-HBc, and positive hepatitis B surface antibody [anti-HBs]) or vaccination (defined as negative HBsAg, negative anti-HBc, and positive anti-HBs) may be eligible to participate.
* Has history of immune suppression disorders
* Has received a live (attenuated) vaccine within the last 60 days, including subjects who plan to receive live (attenuated) vaccines during the study or within 60 days after the final dose of study treatment.
* Has received influenza vaccine within 14 days of screening.
* Has received a biologic or immunotherapy in the last 6 months (If receiving allergy shots with stable dosing, is acceptable)
* Has received prescription or non-prescription medication and in the opinion of the Investigator, the product will interfere with the study procedures or data integrity or compromise the safety of the subject.
* Subjects with clinically significant abnormal laboratory test values in screening blood samples. In particular subjects with the following should be excluded:

Subjects with abnormal coagulation panel at screening such as abnormal PT or aPTT or fibrinogen

Abnormal liver function tests:

Liver enzyme abnormalities (except in the case of known Gilbert's syndrome)

AST or ALT ≥3x ULN and total bilirubin ≥2x ULN AST or ALT ≥5x ULN AST or ALT ≥3x ULN if associated with appearance or worsening of rash or hepatitis symptoms Abnormal platelet counts (<150,000/mcL or > 450,000/mcL) Abnormal white blood cell counts (<3E3/uL or > 11E3/uL ) Abnormal eGFR (<60 mL/min/1.73m2) Elevated IgE level above 50 IU/mL

* Subjects planning to undergo Elective procedures or surgeries at any time after signing the ICF through the follow-up visit.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* Recent history of bleeding or bleeding disorders or any condition whereby in the opinion of the treating investigator giving anti-coagulation during treatment would be contraindicated.
* History of hypersensitivity to antihistamines.
* Weight is over 350lbs.
* Subjects with active drug or alcohol abuse within 1 year prior to screening
* Subject is participating in a clinical trial of another investigational drug or device, including subjects who have participated in another study for a duration of 5 half-lives of the investigational agent.
* Investigators could exclude subjects with any medical condition, including, but not limited to, cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, renal, or a psychiatric condition that, in the opinion of the Investigator, could compromise the participant's ability to participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 21 days
  Incidence of abnormal vital signs and abnormal laboratory values
Rate and type of adverse events during and after infusion of OPT101 or placebo | 48 hours
  Collection of all adverse events
Incidence of vital signs | 48 hours
  Continuous telemetry monitoring
Incidence of abnormal laboratory values | 21 days
  Blood laboratory results and iStat results onsite
Definition of maximum tolerated (MTD) single and repeated doses of OPT101 | 48 hours
  DMC and Safety and Tolerability

SECONDARY OUTCOMES:
Determine pharmacokinetic (PK) Parameters (AUC0-t, Cmax, CL/F, t1/2) | 8 hours
  PK samples will be taken at 8 time points during the infusion
Development of anti-drug antibodies after 1 or more infusions | 2 weeks- 1 prior to infusion and day 15
  Anti-drug antibodies will be collected 2 times during study

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Melamed, MD, Principal Investigator — IMMUNOe Health Centers
Locations (1):
- IMMUNOe Research, Centennial, Colorado, United States

IPD SHARING:
Plan to Share IPD: No